CLINICAL TRIAL: NCT06912139
Title: Topical Nitroglycerin Pretreatment for the Prevention of Radial Arterial Spasm
Brief Title: Topical Nitroglycerine for Prevention of Radial Artery Spasm
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other)
Responsible Party: Principal Investigator, Basaraba Gabriela Lavinia, Legal entity appointed representative, University of Medicine and Pharmacy "Victor Babes" Timisoara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11/10.03.2023
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Radial Artery Spasm
Keywords: topical nitroglycerine; radial artery spasm; coronary angiography; radial puncture

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- nitroglycerin topic cream for radial artery spasm prevention, applied before radial artery puncture (Active Comparator)
  Interventions: Drug: Nitroglycerin transdermal
- placebo cream administration (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nitroglycerin transdermal — Nitroglycerin cream is applied ~ 15 minutes before radial artery puncture for emergency or planned invasive cardiology procedure (example: coronary angiography), and radial artery spasm and diameter are determined by angiography, injecting contrast into the radial artery through the placed radial sheath.
  Arms: nitroglycerin topic cream for radial artery spasm prevention, applied before radial artery puncture
Other: Placebo — Placebo cream with no active compounds is applied by the designated nurse to the radial puncture site, similar to NTG cream, with both patient and invasive cardiologist blinded wo which arm the patient is included in.
  Arms: placebo cream administration

SUMMARY:
In a randomized, double-blind trial, 100 patients undergoing angiography were pre-treated with either topical nitroglycerin (NTG) or placebo. Outcomes assessed included radial artery spam (RAS) incidence, radial artery puncture success, number of attempts, procedural duration, patient discomfort, and complications. RAS was evaluated angiographically and clinically, with additional subgroup analyses for diabetic and smoking patients

DETAILED DESCRIPTION:
During the period of April 2023 - June 2023, 100 consecutive patients that un-derwent invasive angiography using radial artery approach (deemed suitable access site by operating physician) were enrolled and randomized to either pretreatment with a topical cream 0.2% NTG, or application of a gel that contained no active substances. Randomization was done using a computer program designed to randomly produce either the digit 1 or 0, with 1 meaning the patient was assigned to nitroglycerine cohort and 0 to placebo cohort. The assigned nurse that handled the randomization also ad-ministered the patient's treatment. The NTG or placebo cream was applied 20-40 minutes before radial artery puncture by the assigned nurse. The study was designed as a randomized, double-blinded trial, with neither the patient nor the operator aware of the treatment allocation. Patients had indication of either elective or emergency coronary artery or peripheral artery angiography, and had no contraindication to ra-dial artery approach. Both right and left radial arteries were used, depending on oper-ator judgement, while distal radial approach was not utilized in any case. The operator assessed the radial artery pulse quality by manual palpation before puncture. Standard local subcutaneous anesthesia with 5 ml of 2% lidocaine solution was performed. A visual analog scale was used to judge patient discomfort related to the puncture and puncture site at several times during the procedure, with the worst pain level being documented (scale of 0 to 10, where 0 is no pain, and 10 is worst possible pain). The key objective was assessing spasm of the radial artery, which was judged both subjectively by the operator by judging the grade of resistance felt during manipulation of the catheters, and objectively by injection of contrast dye into the radial artery through the introducer sheath immediately after it had been placed inside the radial artery. Spasm was defined as narrowing of the radial artery lumen by more than 50%. Diffuse spasm was defined as spasm of a segment of radial artery greater than 2 cm, or more than two different sites of spasm. The diameter of the radial artery was also measured on the radial angiograms, and was indexed to the patient's body surface area. After sheath insertion and radial artery measurement, the operator could administer intraarterial NTG at his discretion throughout the procedure.

Other data that was included was number of attempts that lead to successful puncture and sheath placement, procedure duration (including angioplasty if needed), contrast dye used and hospital stay duration. Patients were screened for cardiovascu-lar risk factors such as smoking, diabetes mellitus, dyslipidemia, hypertension and obesity. Procedural anticoagulation was performed using 5000 units of unfractioned heparin for diagnostic procedures and 70 units/kilogram for angioplasties. At the end of the procedure, after sheath extraction, hemostasis was achieved using a compres-sive dressing that was left in place for ~12 hours. Bleeding complications at the site of puncture were noted (presence of local hematoma), and ultrasound screening at dis-charge was used to check postprocedural radial artery patency.

Radial sheaths used were 6 French, and the operator had the freedom to use any size of catheters he considered, most often choosing 6 French for both diagnostic angi-ography and percutaneous intervention. No preprocedural patient sedation was used, and cath lab temperature was similar for all cases.

Statistical analysis was performed using IBM SPSS Statistics version 20.0 software for Windows with a significant p<0.05. We used descriptive statistics, figures, and ta-bles to summarize our findings. Results for targeted variables were presented using descriptive statistics (mean, standard deviation, range, median, and associated inter-quartile range) for continuous data, and counts with associated percentages for cate-gorical data. Independent samples t-test was used to analyze differences in means for continuous variables, while differences between categorical variables were examined by Chi-squared test. Categorical data are presented as counts (percentages).

ELIGIBILITY:
Inclusion Criteria:

* indication for invasive cardiology procedure (diagnostic or curative)
* deemed suitable for radial access by operating physician

Exclusion Criteria:

* refuses or unable to give consent
* demed unsuitable for radial artery access (no radial pulse, small patient size, anticipation of complex procedure that requires alternative access site)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Radial artery spasm as determined by angiography of radial artery; spasm being defined as >50% stenosis | Baseline

SECONDARY OUTCOMES:
Number of radial artery puncture attempts | Baseline
  Nitroglycerin cream is applied ~15 minutes before radial puncture is attempted, operator notes number of tries to successfully puncture it and place the sheath
Crossover to alternative puncture site | Baseline
  If radial puncture is unsuccessful another puncture site is needed, this is noted by operator as need for cross-over
Radial artery diameter, absolute value | Baseline
  Angiographical measurement of radial artery diameter in non-spastic area
Patient discomfort measured using a Visual Analog Scale | Intraprocedural, every 15 minutes
  The patient is asked throughout the procedure level of pain on a 0-10 scale, and maximum level is noted
Radial artery spasm: diffuse or localized | Baseline
  If radial spasm is present on a segment of radial artery longer than 20mm it is noted as diffuse, if shorter then it is noted as localized
Contrast medium used during procedure | At the end of invasive procedure
  Total amount in milliliters l is noted
Invasive procedure duration | at the end of invasive procedure
  Total duration of procedure is noted, from puncture of artery to catheter withdrawal (coronary angiography, angioplasty, other angiographic investigation)
Hospital stay duration | Up to 10 weeks
  Total length of hospitalization is noted (in days)
Number of patients with radial artery patency at discharge | Up to 3 weeks
  Radial artery patency (of punctured artery) is determined by ultrasound analysis on the day of discharge
Local complications at puncture site - hematoma | Up to 3 weeks
  During hospital stay, after procedure is completed, forearm is examined for local hematoma in relation to radial artery puncture site
Radial artery diameter indexed to body surface area | Baseline
  Angiographical measurement of radial artery diameter in non-spastic area indexed to patient body surface area

CONTACTS AND LOCATIONS:
Locations (1):
- Timisoara Institute for Cardiovascular Diseases, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No